CLINICAL TRIAL: NCT06481033
Title: Reducing Suicide-Specific Rumination in Veterans Using Real-time Functional Magnetic Resonance Imaging Neurofeedback
Brief Title: Suicide Specific Rumination in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5132-P
Record Dates: First submitted 2024-06-17; First posted 2024-07-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Depression; Suicide; Mood Disorders
MeSH Terms: conditions — Depression; Suicide; Mood Disorders

STUDY DESIGN:
Intervention Model Description: The goal of this study is to collect feasibility and acceptability data regarding the utility of using real-time functional magnetic resonance imaging neurofeedback in veterans experiencing suicide-specific rumination defined as a "repetitive mental fixation on one's suicidal thoughts and intentions." Veterans will be provided neurofeedback signals from the brain to identify mental strategies for altering brain connectivity to reduce rumination. Pre- and post-treatment assessments of suicide, disability, functional impairment, and quality of life will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real-time fMRI Neurofeedback (Experimental): This is a pilot study to collect feasibility and acceptability data regarding the utility of real-time functional magnetic resonance imaging feedback for veterans experiencing suicide-specific rumination. All study participants will receive the intervention.
  Interventions: Behavioral: Real Time fMRI Neurofeedback

INTERVENTIONS:
Behavioral: Real Time fMRI Neurofeedback — The proposed pilot study is designed to collect feasibility and acceptability data regarding the utility of real-time functional magnetic resonance imaging (rt-fMRI) feedback in reducing suicide-specific rumination in veterans. Fifteen veterans will receive 2 rt-fMRI neurofeedback sessions while attempting to alter connectivity in brain regions that play a role in rumination. Pre- and post-treatment assessments of suicide, disability, functional impairment, and quality of life will be collected.

SUMMARY:
Few treatments target core features of suicidal thoughts and behaviors in Veterans. Real-time functional magnetic resonance imaging neurofeedback can provide information regarding brain activation associated with suicide-specific rumination, defined as a "repetitive mental fixation on one's suicidal thoughts and intentions." The goal of this feasibility study is for Veterans to learn strategies for modulating activity within brain regions that have been demonstrated to contribute to the maintenance of rumination, as they receive neurofeedback feedback signals from the brain.

DETAILED DESCRIPTION:
Suicide is much higher in Veterans compared to non-Veterans and thus remains a major health crisis in the VA, but there are few treatments available that directly target core features of suicidal thoughts and behaviors. Rumination is the strong tendency to engage in self-critical repetitive thinking that is often difficult to interrupt and is associated with suicide attempts and the transition from suicidal ideation to intent above and beyond other suicide risk factors. Meta-analyses indicate that abnormalities in brain regions comprising the "default mode network," which play a role in daydreaming or mind-wandering, contribute to the maintenance of rumination. Although functional magnetic resonance imaging studies have provided key insights into the neurobiology of suicide, there has been little direct impact on clinical care thus far. With the advent of real-time functional magnetic resonance imaging (rt-fMRI) neurofeedback, however, there is now the potential to implement personalized strategies for altering brain activity associated with rumination to reduce suicidal thoughts and behaviors. In the proposed study the investigators will determine the acceptability and feasibility of using rt-fMRI neurofeedback to reduce suicide-specific rumination, defined as "repetitive mental fixation on one's suicidal thoughts and intentions" in a transdiagnostic sample of 15 Veterans at elevated risk of suicide. The investigators will also assess pre- to post-treatment changes in measures of suicide-specific rumination, disability, functional impairment, and quality of life in Veterans with a suicide attempt history following 2 rt-fMRI neurofeedback sessions. Veterans will be provided signals from the brain to identify mental strategies (e.g., cognitive reappraisal) for altering brain connectivity. During a subsequent "transfer" period Veterans will be asked to utilize the mental strategy that worked best for altering this connectivity, but without receiving any neurofeedback signals from the brain. Post-treatment clinical assessments will occur following each of the 2 rt-fMRI neurofeedback sessions and at 1 month following the second fMRI neurofeedback session. The novelty of the proposed work is underscored by the paucity of work using rt-fMRI neurofeedback in a Veteran population and the lack of studies to date targeting a brain network to reduce suicide-specific rumination. In this study the investigators will test the following specific aims: (1) to determine the acceptability and feasibility of implementing rt-fMRI neurofeedback in a Veteran population experiencing suicide-specific rumination; (2) to identify changes in suicide-specific rumination following rt-fMRI neurofeedback and (3) to identify changes in functional impairment and quality of life following rt-fMRI neurofeedback. The proposed study is consistent with the mission of RR&D to maximize Veterans' functional independence, quality of life and participation in their lives and community.

ELIGIBILITY:
Inclusion Criteria:

* U.S. military veteran between 18-65 years old
* negative pregnancy test on MRI scan days
* score greater than or equal to 10 on the Suicide Rumination Scale
* clinically stabilized on psychotropic medications
* engaged in mental health care treatment
* able to provide written, informed consent

Exclusion Criteria:

* no major medical or neurological disorders that could interfere with treatment
* moderate or severe traumatic brain injury
* current imminent suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the assessor
* any current psychotic disorder
* MRI contraindications
* any substance use disorder for substances other than cannabis or alcohol (mild alcohol or cannabis use disorder does not exclude participants but moderate or severe alcohol or cannabis substance use disorder is disqualifying)
* pregnant or trying to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability and Feasibility | Total score obtained 2 weeks following first real-time fMRI neurofeedback session.
  The Client Satisfaction Questionnaire will be used to assess acceptability and feasibility of implementing real-time fMRI neurofeedback in a Veteran population. The total score on the questionnaire ranges from from 8 to 32 with higher scores indicative of greater satisfaction.

SECONDARY OUTCOMES:
Suicide Rumination Scale | Change in total score from pre-treatment to post-treatment (2 weeks).
  The Suicide Rumination Scale is a self-report inventory designed to quantify the extent to which an individual ruminates about suicide. The total score on the scale ranges from 0 to 32 with higher scores indicative of greater rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Szeszko, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will obtain IRB approval prior to sharing de-identified data.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared with scientific collaborators after the data have been analyzed and submitted for publication.
Access Criteria: De-identified data will be shared when the study is completed and following IRB approval.